CLINICAL TRIAL: NCT04479696
Title: Novel Intervention to Reduce Patient and Caregiver Anxiety Around Radiation Treatment for Brain Tumors With a Customized Neuro-Imaging Referenced Symptom Video
Brief Title: Customized Neuro-Imaging Referenced Symptom Video for the Reduction of Patient and Caregiver Anxiety Around Radiation Treatment for Brain Tumors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018-0097; NCI-2020-03698 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0097 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-07-16; First posted 2020-07-21 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-01

CONDITIONS: Glioblastoma; WHO Grade II Glioma; WHO Grade III Glioma
MeSH Terms: conditions — Glioblastoma | interventions — Early Intervention, Educational; Educational Status; Methods; Videotape Recording

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (NIRS) (Experimental): Patients receive standard of care verbal and written education materials. Patients also receive a customized video which includes a description of each of their tumor, functional areas of the brain affected, and possible symptoms from the tumor and radiation treatment based on the neuro-imaging features. Patients and their caregivers watch the video together or separately over 1.5-3 minutes before the end of the first week of radiation treatment. Within 2 weeks after watching the NIRS video, patients complete an optional survey over 5-10 minutes.
  Interventions: Other: Educational Intervention; Other: Questionnaire Administration; Other: Survey Administration; Other: Video
- Arm II (standard of care) (Active Comparator): Patients receive standard of care verbal and written education materials.
  Interventions: Other: Educational Intervention; Other: Questionnaire Administration

INTERVENTIONS:
Other: Educational Intervention — Receive standard of care verbal and written education materials
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
Other: Questionnaire Administration — Ancillary studies
Other: Survey Administration — Complete optional survey
  Arms: Arm I (NIRS)
Other: Video — Watch NIRS video
  Arms: Arm I (NIRS)

SUMMARY:
This trial studies whether a customized video intervention can help to reduce anxiety in brain cancer patients undergoing radiation treatment and their caregivers. A customized neuro-imaging referenced symptom video that describes symptoms and side effects specific to the patients' tumor may result in an early and sustained reduction in anxiety and distress during and after radiation treatment, thereby improving quality of life.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine if provision of a neuro-imaging referenced symptom (NIRS) video intervention for patients starting radiotherapy for newly diagnosed primary brain tumors reduces patient anxiety during radiation compared to standard of care information.

SECONDARY OBJECTIVES:

I. To determine if provision of a NIRS video intervention for patients starting radiotherapy for newly diagnosed primary brain tumors reduces caregiver anxiety during radiation compared to standard of care information.

II. To determine if any changes in patient or caregiver anxiety early during radiation are sustained after the completion of radiation.

III. To investigate whether changes in anxiety are associated with changes in quality of life and distress in patients.

IV. To investigate whether patients perceive the NIRS intervention to have been helpful in understanding possible tumor and treatment symptoms.

OUTLINE: Patients and their caregivers are randomized to 1 of 2 arms.

ARM I (NIRS VIDEO): Patients receive standard of care verbal and written education materials. Patients also receive a customized NIRS video which includes a description of each their tumor, functional areas of the brain affected, and possible symptoms from the tumor and radiation treatment based on the neuro-imaging features. Patients and their caregivers watch the video together or separately over 1.5-3 minutes before the end of the first week of radiation treatment. Within 2 weeks after watching the NIRS video, patients complete an optional survey over 5-10 minutes.

ARM II (STANDARD OF CARE EDUCATION): Patients receive standard of care verbal and written education materials.

After completion of radiation treatment, patients are followed up at 1 month.

ELIGIBILITY:
Inclusion Criteria:

* PATIENT ELIGIBILITY CRITERIA: Adult patients with newly diagnosed glioma (World Health Organization [WHO] grade 2-4) who are planned for a 6-week course of radiotherapy after surgery
* PATIENT ELIGIBILITY CRITERIA: Able to complete questionnaires in English
* PATIENT ELIGIBILITY CRITERIA: Has a post-operative diagnostic magnetic resonance imaging (MRI) of the brain with and without contrast acquired within 4 weeks of the start of radiotherapy
* CAREGIVER ELIGIBILITY CRITERIA: Adult caregiver (>= 18 years) who is accompanying an eligible patient consented to the study
* CAREGIVER ELIGIBILITY CRITERIA: The patient who the caregiver is accompanying is consented for participation on the study
* CAREGIVER ELIGIBILITY CRITERIA: Able and willing to complete questionnaires in English

Exclusion Criteria:

* PATIENT ELIGIBILITY CRITERIA: Significant cognitive or psychiatric symptoms that prevent the ability to complete the questionnaires as determined by the assessing staff in the pre-intervention evaluation
* PATIENT ELIGIBILITY CRITERIA: Poor performance status (Karnofsky performance status [KPS] < 60) that prevent the ability to complete the questionnaires
* CAREGIVER ELIGIBILITY CRITERIA: Significant cognitive or psychiatric symptoms that prevent the ability to complete the questionnaires as determined by the assessing staff in the pre-intervention evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 117 (Estimated)
Dates: Start 2019-06-05 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Changes in patient S-Anxiety subscale score of the State-Trait Anxiety Inventory (STAI) | From baseline to 2 weeks, 6 weeks and 1 month post-radiation therapy (RT)
  Using linear mixed models (LMMs) to evaluate the change in STAI between and within groups. The correlation structure over time will be selected using the Bayesian information criterion. Will calculate correlations between reduction in anxiety and improvement in quality of life (Functional Assessment of Cancer Therapy Scale-Brain [FACT- Br]) and distress (Distress Thermometer). Analysis will focus on the between-group comparison of the changes of the patient S-Anxiety subscale score of the STAI from baseline to 2 weeks and from baseline to 6 weeks in to RT. All tests conducted will use a two-sided 0.05 significance level, without adjusting for multiple testing.

SECONDARY OUTCOMES:
Changes in caregiver S-Anxiety subscale score of the STAI and Distress Thermometer score | From baseline to 2 and 6 weeks
  Analysis will focus on the between-group comparison of the changes of the caregiver S-Anxiety subscale score of the STAI from baseline to 2 weeks and from baseline to 6 weeks in to RT. All tests conducted will use a two-sided .05 significance level, without adjusting for multiple testing.
Change in patient and caregiver S-Anxiety subscale score of the STAI and Distress Thermometer scores | From baseline to 1 month post-RT
  Analysis will be performed by testing for the effects of time, in particular, differences between the average of weeks 2 and 6 during RT and 1 month after RT. All tests conducted will use a two-sided .05 significance level, without adjusting for multiple testing.
Changes in patient Distress Thermometer score and FACT-Br score | From baseline to 2 weeks, 6 weeks, and 1 month post-RT
  Evaluates the impact between distress and overall quality of life in patients. LMMs will be used to assess the correlations between change in anxiety and change in quality of life, etc., without including time as an independent variable, yet with within-subject correlations still accounted for. For each fixed time point, simple correlations will also be calculated. All tests conducted will use a two-sided .05 significance level, without adjusting for multiple testing.
Patient survey | Up to 1 month post-RT
  Evaluates whether neuro-imaging referenced symptom intervention was subjectively helpful in understanding their tumor and treatment symptoms and alleviating their anxiety. Relevant summary statistics will be computed. All tests conducted will use a two-sided .05 significance level, without adjusting for multiple testing.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Chung, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org